CLINICAL TRIAL: NCT02088489
Title: Effectiveness and Safety of Porous Tip Irrigated Ablation Catheter Versus Conventional Irrigated Catheter in Isthmus Dependent Atrial Flutter Ablation: a Randomized Study
Brief Title: Thermocool SF Catheter Versus Thermocool Catheter in Isthmus-dependent Atrial Flutter Ablation
Acronym: Cathena
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of the Arrhythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF vs Tc
Record Dates: First submitted 2014-02-26; First posted 2014-03-17 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Atrial Flutter
Keywords: Atrial flutter; Thermocool catheter; Thermocool SF catheter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atrial flutter, irrigated catheter (Active Comparator): Patients with isthmus dependent atrial flutter, undergone to catheter ablation with Thermocool® (Biosense Webster, Diamond Bar, CA) irrigated catheter
  Interventions: Device: Atrial flutter irrigated catheter
- Atrial flutter, porous tip catheter (Experimental): Patients with isthmus dependent atrial flutter, undergone to catheter ablation with Thermocool® SF(Biosense Webster, Diamond Bar, CA) irrigated catheter
  Interventions: Device: Atrial flutter porous tip catheter

INTERVENTIONS:
Device: Atrial flutter irrigated catheter — A duodecapolar isthmic curve catheter will be introduced to demonstrate cavo-tricuspidal bidirectional block. We performed atrial flutter ablation with conventional irrigated Thermocool® (Biosense Webster, Diamond Bar, CA) catheter Continuous lesions from tricuspidal annulus to inferior vena cava will be realized and then complete isthmic block will be confirmed by bidirectional stimulation
  Arms: Atrial flutter, irrigated catheter
Device: Atrial flutter porous tip catheter — A duodecapolar isthmic curve catheter will be introduced to demonstrate cavo-tricuspidal bidirectional block. We performed atrial flutter ablation with Porous tip Thermocool® SF(Biosense Webster, Diamond Bar, CA)irrigated catheter Continuous lesions from tricuspidal annulus to inferior vena cava will be realized and then complete isthmic block will be confirmed by bidirectional stimulation
  Arms: Atrial flutter, porous tip catheter

SUMMARY:
Porous tip catheter use reduces procedure time and RF time in atrial flutter ablation with the same safety.

DETAILED DESCRIPTION:
New porous tip catheters appear more effective in atrial fibrillation ablation than conventional irrigated catheter, with the same safety. We could hypothesize porous tip irrigated catheters are more effective than conventional irrigated catheter, reducing procedure time and RF ablation time.We realize a randomized comparison study.

For that, 70 patients with an indication for isthmus-dependent atrial flutter ablation will be randomized to conventional irrigated catheter ablation or porous tip irrigated catheter ablation. A ECG-Holter examination will be done at 1 month follow up after catheter ablation, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergone to cti-dependent atrial flutter ablation.

Exclusion Criteria:

* Left atrial flutter or atrial fibrillation
* Femoral venous access not available.
* Anticoagulation not therapeutic in patients at high thrombo-embolic risk
* Other contraindications to radiofrequency ablations: pregnancy, malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Time needed to block cavo-tricuspidal isthmus | During ablation procedure

SECONDARY OUTCOMES:
Radiofrequency time. | During ablation procedure
  Total radiofrequency time needed to achieve cavo-tricuspidus isthmus (CTI) block.
Fluoroscopy time. | During ablation procedure.
  Total X-ray time needed to achieve CTI block.
Complications during the procedure. | During ablation procedure.
Survival free from flutter | Up to 12 months after procedure.
  Proportion of patients not presenting with an atrial flutter recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Mont, MD, PhD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Cosio FG, Lopez-Gil M, Goicolea A, Arribas F, Barroso JL. Radiofrequency ablation of the inferior vena cava-tricuspid valve isthmus in common atrial flutter. Am J Cardiol. 1993 Mar 15;71(8):705-9. doi: 10.1016/0002-9149(93)91014-9. PMID 8447269
- [Background] Ilg KJ, Kuhne M, Crawford T, Chugh A, Jongnarangsin K, Good E, Pelosi F Jr, Bogun F, Morady F, Oral H. Randomized comparison of cavotricuspid isthmus ablation for atrial flutter using an open irrigation-tip versus a large-tip radiofrequency ablation catheter. J Cardiovasc Electrophysiol. 2011 Sep;22(9):1007-12. doi: 10.1111/j.1540-8167.2011.02045.x. Epub 2011 Mar 31. PMID 21453368
- [Background] Cuesta A, Mont L, Alvarenga N, Rogel U, Brugada J. Comparison of 8-mm-tip and irrigated-tip catheters in the ablation of isthmus-dependent atrial flutter: a prospective randomized trial. Rev Esp Cardiol. 2009 Jul;62(7):750-6. doi: 10.1016/s1885-5857(09)72355-2. English, Spanish. PMID 19709510
- [Background] Scaglione M, Blandino A, Raimondo C, Caponi D, Di Donna P, Toso E, Ebrille E, Cesarani F, Ferrarese E, Gaita F. Impact of ablation catheter irrigation design on silent cerebral embolism after radiofrequency catheter ablation of atrial fibrillation: results from a pilot study. J Cardiovasc Electrophysiol. 2012 Aug;23(8):801-5. doi: 10.1111/j.1540-8167.2012.02298.x. Epub 2012 Apr 11. PMID 22494043
- [Background] Dixit S, Gerstenfeld EP, Callans DJ, Cooper JM, Lin D, Russo AM, Verdino RJ, Patel VV, Kimmel SE, Ratcliffe SJ, Hsia HH, Nayak HM, Zado E, Ren JF, Marchlinski FE. Comparison of cool tip versus 8-mm tip catheter in achieving electrical isolation of pulmonary veins for long-term control of atrial fibrillation: a prospective randomized pilot study. J Cardiovasc Electrophysiol. 2006 Oct;17(10):1074-9. doi: 10.1111/j.1540-8167.2006.00558.x. Epub 2006 Jul 18. PMID 16879626
- [Background] Feld GK, Fleck RP, Chen PS, Boyce K, Bahnson TD, Stein JB, Calisi CM, Ibarra M. Radiofrequency catheter ablation for the treatment of human type 1 atrial flutter. Identification of a critical zone in the reentrant circuit by endocardial mapping techniques. Circulation. 1992 Oct;86(4):1233-40. doi: 10.1161/01.cir.86.4.1233. PMID 1394929
- [Background] Fischer B, Haissaguerre M, Garrigues S, Poquet F, Gencel L, Clementy J, Marcus FI. Radiofrequency catheter ablation of common atrial flutter in 80 patients. J Am Coll Cardiol. 1995 May;25(6):1365-72. doi: 10.1016/0735-1097(95)00029-4. PMID 7722135
- [Background] Scavee C, Jais P, Hsu LF, Sanders P, Hocini M, Weerasooriya R, Macle L, Raybaud F, Clementy J, Haissaguerre M. Prospective randomised comparison of irrigated-tip and large-tip catheter ablation of cavotricuspid isthmus-dependent atrial flutter. Eur Heart J. 2004 Jun;25(11):963-9. doi: 10.1016/j.ehj.2004.03.017. PMID 15172468
- [Background] McGreevy KS, Hummel JP, Jiangang Z, Haines DE. Comparison of a saline irrigated cooled-tip catheter to large electrode catheters with single and multiple temperature sensors for creation of large radiofrequency lesions. J Interv Card Electrophysiol. 2005 Dec;14(3):139-45. doi: 10.1007/s10840-006-5635-1. Epub 2006 Jan 18. PMID 16421689